CLINICAL TRIAL: NCT04867356
Title: Effects Of Latissimus Dorsi Stretching On Functional Disability Related To Chronic Low Back Pain
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Health Education Research Foundation (HERF) (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: HERF/REC/2021-1
Record Dates: First submitted 2021-04-27; First posted 2021-04-30 (Actual); Last update posted 2021-07-07 (Actual); Status verified 2021-07

CONDITIONS: Mechanical Low Back Pain
MeSH Terms: conditions — Low Back Pain

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Spinal Stabilization Exercises (SSE) (Active Comparator)
  Interventions: Other: Spinal Stabilization Exercises (SSE)
- Spinal Stabilization Exercises (SSE) & Latissimus Dorsi Stretching (LDS) (Experimental)
  Interventions: Other: Spinal Stabilization Exercises (SSE) & Latissimus Dorsi Stretching (LDS)

INTERVENTIONS:
Other: Spinal Stabilization Exercises (SSE) — Spinal stabilization exercises (SSE) including bridging, planks and tummy tuck-in will be performed. Each participant received a total 7 session thrice a week sessions in two weeks, . Each session had lasted for 30-40 minutes. Spinal stabilization exercises were repeated 5-15 times depending on the endurance of patients.
  Home exercise plan will also be given e.g. postural care, precautions in lifting and carrying weights etc.
  Arms: Spinal Stabilization Exercises (SSE)
Other: Spinal Stabilization Exercises (SSE) & Latissimus Dorsi Stretching (LDS) — In experimental group in addition SSE group interventions, participants will receive the latissimus dorsi stretching (LDS). Each participant received a total 7 session thrice a week sessions in two weeks. Each session had lasted for 30-40 minutes. each stretch of latissimus dorsi was of 20-30 seconds with 10-20 repetitions in each session.
  Arms: Spinal Stabilization Exercises (SSE) & Latissimus Dorsi Stretching (LDS)

SUMMARY:
The main objective of the study is to determine effects of latissimus dorsi stretching on functional disability related to chronic low back pain

DETAILED DESCRIPTION:
A single-blinded,randomized clinical trial will be conducted in /multiple rehabilitation centers of Rawalpindi and Islamabad, after taking approval from ERB/IRB respective centers. The study duration will be 3 months. the study participants will be having mechanical low back pain.

The intervention will be included latissmus dorsi stretching along with spinal stabilization exercises in one group and in comparative group spinal stabilization exercises alone. Oswestry Disability Index (ODI) will be used to measure the disability related to the chronic low back pain.

ELIGIBILITY:
Inclusion Criteria:

* male and female
* 20 to 60 years
* chronic mechanical low back pain

Exclusion Criteria:

* patients who had any type of injury or fracture which limits rehabilitation
* patients with the symptoms of radiating pain
* who had disc pathology and spinal cord injury
* patients with medical conditions

Ages: 20 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 61 (Actual)
Dates: Start 2021-01-01 (Actual); Primary Completion 2021-05-30 (Actual); Study Completion 2021-06-01 (Actual)

PRIMARY OUTCOMES:
Oswestry disability index | 2 weeks
  The Oswestry Disability Index (aka the Oswestry Low Back Pain Disability Questionnaire) is an extremely important tool that researchers and disability evaluators use to measure a patient's permanent functional disability. The test has been around since 1980 and is considered the 'gold standard' of low back pain functional outcome tools. SCORE DISABILITY LEVEL 0 - 4 No disability 5 - 14 Mild disability 15 - 24 Moderate disability 25 - 34 Severe disability 35 - 50 Completely disabled The Oswestry Disability Index (aka the Oswestry Low Back Pain Disability Questionnaire) is an ex- tremely important tool that researchers and disability evaluators use

CONTACTS AND LOCATIONS:
Locations (1):
- NOSIS clinics Mansehra Pakistan, Mānsehra, Pakistan

IPD SHARING:
Plan to Share IPD: Undecided